CLINICAL TRIAL: NCT03727386
Title: A Study Evaluating the Feasibility of Undertaking an Intervention Looking Into the Effect of Vegetable Oils Intake on Cognition and Quality of Life in Adults With Mild Cognitive Impairment.
Brief Title: The Effect of Vegetable Oil on Cognitive Functions of MCI Patients
Acronym: DICe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bournemouth University (Other)
Collaborators: Dorset HealthCare University NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1718/IRASREZ/1
Record Dates: First submitted 2018-07-13; First posted 2018-11-01 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Metabolic Ketosis; Cognitive Impairments, Mild
MeSH Terms: conditions — Ketosis; Cognitive Dysfunction | interventions — Coconut Oil; Sunflower Oil

STUDY DESIGN:
Intervention Model Description: This study will be a pilot study with an internal feasibility study that aims at evaluating the acceptance and adherence of participants to the intervention. Participants will be randomized into an intervention (coconut oil) and control group (sunflower oil) using an online randomisation software; Sealed envelope.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coconut oil (Experimental): A dietary intervention that relies on the administration of 30 ml of extra virgin coconut oil per day for six months will be utilized in this study. Coconut oil administered will replace the cooking/vegetable oil usually used by the participants. .
  Interventions: Other: Coconut oil
- Sunflower oil (Placebo Comparator): A dietary intervention that relies on the administration of 30 ml of sunflower oil per day for 6 months will be utilized in this study. The oil administered will replace the cooking/vegetable oil usually used by the participants.
  Interventions: Other: Sunflower oil

INTERVENTIONS:
Other: Coconut oil — Participants will receive 30 ml of virgin coconut oil to replace their normal oil intake for a period of 6 months.
  Other Names: extra virgin coconut oil
  Arms: Coconut oil
Other: Sunflower oil — Participants will receive 30 ml of sunflower oil to replace their normal oil intake for a period of 6 months.
  Arms: Sunflower oil

SUMMARY:
This study explores the feasibility of applying an intervention using vegetable oils (coconut and sunflower oils) on individuals diagnosed with Mild Cognitive Impairment. Participants will be divided into two groups and will either receive 30 ml of coconut or sunflower oil to be consumed daily for six months.

DETAILED DESCRIPTION:
Research has shown that some forms of dementia associated to ageing can often be linked to low levels of sugar in the brain. Which may cause damage to the brain nerve cells. The main source of fuel for the brain comes from sugar in the form of glucose. Providing an additional source of fuel to brain cells may reduce the damage, potentially preventing further decline of dementia in individuals with Mild Cognitive Impairment (MCI).

This study explores the possibility of using vegetable oils (coconut and sunflower oils) as an additional source of energy to individuals diagnosed with Mild Cognitive Impairment. The researchers will use different tests to evaluate if the study could be done. Participants will be divided into two groups and will either receive 30 ml of coconut or sunflower oil to be consumed daily for six months. The researchers will visit participants in their houses over three times during the study to collect the data.

During each visit, the researcher will conduct blood test in which blood will be collected by pricking the finger of participants to check their blood ketone levels. Paper pencil and/or computer tasks will be completed to measure the cognitive abilities (e.g. attention, orientation and learning) of participants. Participants will also be asked to complete a food diary in which they will provide details of their diet and eating habits. Moreover, they will be asked to provide feedback on the study by answering a set of questions either during an interview or by completing a feedback form. The information collected during these visits will be used to evaluate the study.

Results from this study would help determine whether such an intervention can be undertaken in adults with MCI. The study will provide information related to the practicality of using vegetable oils on adults with MCI. This would provide the evidence to develop a larger study that would allow us to systematically evaluate the effect of vegetable oils on MCI. Which would further enable us to develop an intervention that might possibly improve the brain functions of adults with MCI and maintain their quality of life for longer by delaying the development of dementia and reducing the progression from MCI to AD (Alzheimer's disease) in adults.

ELIGIBILITY:
Inclusion Criteria:

* Adults with confirmed MCI diagnosis
* Adults with Negative Apo E4 genotype

Exclusion Criteria:

* Adults diagnosed with Alzheimer's Disease (AD)
* Adults with positive Apo E4 genotype
* Adults with confirmed diabetes (Type I, Type II) diagnosis
* Adults with a history of hyper-cholesterolemia (high cholesterol levels) or Dyslipidaemia
* Adults who are unable to understand written or verbal English
* Adults diagnosed with Neurological disorders (Parkinson, stroke…)
* Adults with post traumatic brain injury (tumour, brain surgery, injury…)
* Patients with major physical impairments (blind, deaf) or those who are unable to use their dominant hand.
* Adults with coconut allergy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-11-19 (Actual); Primary Completion 2021-05-06 (Actual); Study Completion 2021-05-06 (Actual)

PRIMARY OUTCOMES:
Vegetable oil usage | 6 months
  the amount of oil used by individuals (ml) will be monitored

SECONDARY OUTCOMES:
Overall cognition | Six months
  Assessed by Mini Addenbrookes Cognitive Examination (mACE) which has a high score of 30 with higher scores indicating better cognition.
Quality of life of adults with Mild cognitive impairment measured by ADCS-MCI-ADL (Alzheimer's Disease Cooperative Study Mild Cognitive Impairment- Activities of Daily Living) | six months
  Quality of life of participants measured by ADCS-MCI-ADL (Alzheimer's Disease Cooperative Study Mild Cognitive Impairment- Activities of Daily Living) questionnaire, it has a score that rages from 0 to 53; higher score are linked to better quality of life.
Dietary intake assessed by four day food records using Nutritics software | six months
  Dietary energy and macronutrient (carbohydrate, fat and protein) intake assessed by four day food records using Nutritics software (https://www.nutritics.com/p/references).
Blood samples (beta hydroxyl butyrate): | six months
  ketone bodies concentrations (mmol) will be assessed by Abbott freestyle Optium Neo, ketone meter.
Executive measure | six months
  Assessed by trail making test B that has an average score of 75 seconds and a deficient score of > 273 seconds
Verbal Memory | six months
  Verbal memory will be assessed by word list test which is a subtest of the Wechsler Memory Scale III; the lower the test score the higher the cognitive impairment.
Verbal Fluency | six months
  Verbal Fluency test in which a score lower than 17 shows cognitive impairment (the higher the score the better the cognition) will be used to determine
Processing Speed | six months
  Digit symbol test in which lower test scores are correlated with higher impairment will be used to assess processing speed
Attention | six months
  Digit Span test will be used to assess attention, the lower the score the higher the impairment.
Visual Spatial memory | six months
  Supermarket task will be used to asses the visual spatial memory of participants, the score depends on the time required to complete the task. Extra time is related to higher cognitive impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Raysa EL Zein, MSc, Principal Investigator — Student; Jane Murphy Professor, PhD, Study Director — Professor of Nutrition; Peter Thomas Professor, PhD, Study Director — Professor of Health Care Stats & Epidemiology; Shanti Shanker Doctor, PhD, Study Director — Lucturer of Psychology
Locations (1):
- Bournemouth University, Bournemouth, Dorset, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers.